CLINICAL TRIAL: NCT03272971
Title: Feasibility Study of the RF Ablation Catheter to Ablate Lung Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Broncus Medical Inc (Industry)
Collaborators: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Protocol 45
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Lung Cancer, Non-small Cell
Keywords: lung cancer; radiofrequency ablation; bronchoscopy; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Radio-frequency Ablation (Experimental): Single-arm study where subjects receive radio-frequency ablation prior to a scheduled, surgical resection.
  Interventions: Device: Radio-frequency Ablation

INTERVENTIONS:
Device: Radio-frequency Ablation — The intervention consists of a bronchoscopic approach to ablate lung tumors with radiofrequency.

SUMMARY:
The feasibility of a RF ablation catheter to bronchoscopically ablate lung tumors, will be evaluated in patients already scheduled for surgical resection.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center, pilot study of bronchoscopic Radio-Frequency Ablation (RFA) treatment of target lung lesions, prior to surgical tumor resection. Up to ten (10) subjects will be treated at the investigational site.

Subjects identified for this study will be those that have a surgical resection already scheduled as part of their lung cancer treatment. Patients who have consented to participate in this study (enrolled) will undergo screening assessments to evaluate the inclusion criteria associated with their lung cancer and general health. Only patients that meet all of the inclusion criteria and none of the exclusion criteria will be scheduled for RFA treatment.

Prior to RFA, high-resolution computed tomography (HRCT) scans will be used to characterize the lesion and determine the access pathways for ablation. At the time of the RFA procedure, a point-of-entry, along a bronchial wall, is created under an image-guided navigation system. The RFA catheter is advanced down the access path until it reaches the tumor and RF is administered at the prescribed dose. Upon completion of the RFA treatment, the subject is immediately prepared for surgical resection in accordance with their lung cancer standard of care. There are no follow-up visits as part of this study, the subject is excited following surgical resection.

The resected tissue will undergo pathological evaluation for tissue viability.

ELIGIBILITY:
Inclusion Criteria:

* Proven NSCLC or pulmonary metastases from extra-thoracic primary tumor
* Must be eligible for curative lung resection (lobectomy)
* Tumor/lesion size will be a minimum of 10mm along the minor diameter
* Willing to participate in all aspects of study protocol for duration of the study
* Able to understand study requirements
* Signs informed consent form

Exclusion Criteria:

* Any contraindication to bronchoscopy, for example:

  * Untreatable life-threatening arrhythmias.
  * Inability to adequately oxygenate the patient during the procedure.
  * Acute respiratory failure with hypercapnia (unless the patient is intubated and ventilated).
  * Recent myocardial infarction.
  * Previously diagnosed high-grade tracheal obstruction.
  * Uncorrectable coagulopathy
* Known coagulopathy
* Platelet dysfunction or platelet count <100 x 10^3 cells/mm3
* History of major bleeding with bronchoscopy
* Suspected pulmonary hypertension: additional testing required, such as ECG
* Moderate-to-severe pulmonary fibrosis
* Severe emphysema (GOLD III/IV) or chronic obstructive pulmonary disease (COPD):

additional testing and PI consent is required

* Bullae >5cm located within the same lobe of target tumor/lesion
* Any other severe or life-threatening comorbidity that could increase the risk associated with bronchoscopic RFA
* Ongoing systemic infection
* Contraindications to general anesthesia
* Inability to stop anticoagulants or antiplatelet agents prior to procedure as dictated by the protocol
* Prior thoracic surgery on the same side of the lung as the targeted tumor/lesion
* Breastfeeding women or females of childbearing potential with a positive pregnancy test prior to the procedure or the intent to become pregnant during the study
* Life expectancy of less than one year.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
RFA relate AEs/SAEs | Day 0
  The incidence of reported adverse events and serious adverse events related to the RFA procedure
Feasibility - Ablated Tissue | Day 0
  Semi-quantitative scoring of necrotic tissue assessed by histology
Feasibility - Delivery of Ablation | Day 0
  Treatment meets the required procedural steps/requirements per the Operator's Manual and treatment is delivered to the target tumor per the individual patient navigation plan.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China